CLINICAL TRIAL: NCT01077388
Title: Collaborative Behavioral e-Care to Decrease Cardiovascular Risk (e-Compare)
Brief Title: e-Care for Heart Wellness
Acronym: e-Compare
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2R01HL075263-05 (NIH)
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: CVD
Keywords: CVD; uncontrolled HTN

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietician electronic counseling (Experimental): This arm will receive care and supportive emails and phone calls from a study dietician for about 6 months. We will also provide a blood pressure monitor, a pedometer, and a scale with instructions for using them at home.
  Interventions: Behavioral: Dietician electronic support
- Self Care (No Intervention): This arm will continue to get care as usual from their regular doctor. They will also get a blood pressure monitor and a scale at the end of the study.

INTERVENTIONS:
Behavioral: Dietician electronic support — Dietitian-delivered behavioral intervention, that uses a patient shared EMR and e-communications, will be integrated into routine healthcare and will result in improved control of modifiable CVD risk.
  Arms: Dietician electronic counseling

SUMMARY:
The e-Care for Heart Wellness study will look at ways to reduce a person's chances of getting heart disease. We are asking about 100 Group Health members whose electronic medical record shows they have uncontrolled high blood pressure to be in the study. Having high blood pressure increases your future risk of heart attacks and strokes.

There are many things you can do to help keep your heart healthy. Examples include lowering blood pressure and cholesterol, eating healthier, and being more active. Our goal is to test whether getting care and supportive emails from a dietician helps people do things like this to lower their chances of having a heart attack or a stroke.

For some people, this study will involve both research and clinical care. About half the people in the study will receive care related to heart disease prevention from a dietician. It's a standard clinical practice for dieticians to help people reduce their risk of heart attacks and strokes. What's different about this study is using emails from a dietician to help people take steps to improve their heart health.

DETAILED DESCRIPTION:
Overweight and obese adults are more likely to have hypertension and other risk factors for cardiovascular disease (CVD). Evidence-based medication and lifestyle strategies exist for reducing CVD risk, but little is known about the comparative effectiveness and cost-effectiveness of these strategies and how best to integrate them into routine health care. We have previously demonstrated that Web-based pharmacist medication management intervention can cost-effectively improve HTN control (e-BP: Electronic Communication and Home Blood Pressure Monitoring; R01 HL075263, B. Green, PI). Web-based pharmacy care did not lead to lifestyle behavior change or weight loss. However patients who lost small amounts of weight (2 kg or more) were more likely to have controlled BP (p=.008), regardless of their study group assignment. We propose using Health Information Technology systems (HIT) to identify asymptomatic patients at moderate risk for CVD and invite them to participate in a theory-based behavioral intervention that uses the Chronic Care Model as its planning foundation.

Specific Aims Aim #1: We hypothesize that using electronic databases alone, we can identify asymptomatic overweight or obese patients, with uncontrolled BP, and at moderate risk for CVD who might benefit from a behavioral intervention.

Aim #2: We hypothesize that a dietitian-delivered behavioral intervention, that uses a patient shared EMR and e-communications, can be integrated into routine healthcare and will result in improved control of modifiable CVD risk. To test this hypothesis we will measure:

Primary outcomes:

1. The proportion of patients who agree to participate and complete the intervention.
2. The change in mean systolic and diastolic BP and weight (kg), and a weight loss of 4 kg or more, and the change in Framingham risk score.

Secondary outcomes:

1. Patient satisfaction with the intervention, its effects on health related quality of life (HrQOL) and the cost of delivering the intervention.

Using this information and the results of the e-BP trial we will plan a full scale, multi-site (2-3 health institutions with comprehensive EMR's and different geographic and patient populations) multi-factorial randomized trial-to test the comparative effectiveness of different strategies to improve control of modifiable CVD risk.

ELIGIBILITY:
Inclusion Criteria:

* All adults age 30-<70 men and women who have received care at GH primary care medical centers in Western Washington and who have been continuously enrolled in GH for at least 2 years.
* BMI 26 or higher,
* Uncontrolled HTN (based on the 2 most recent visits), and moderate risk for CVD.

Exclusion Criteria:

* A history of any type of cardiovascular disease (CVD). Including TIA, stroke, coronary heart disease (CHD), angina, congestive heart failure (CHF), peripheral arterial disease (PAD), ar, CHF, PAD), arrhythmias, cardiomyopathy, and valvular disease.
* Pre existing diagnosis of diabetes
* Diagnosis of a serious life threatening or limiting condition
* Pre existing diagnosis of alcohol or chemical dependency
* Pregnant or planning on becoming pregnant in the next 6 months. Women randomized to the intervention group who become pregnant during the study will be given the option of continuing the intervention in conjunction with usual pre-natal care provided by GH, but will not be included in the final analysis for the study. Women randomized to the self care group who become pregnant during the study will be given the home monitoring equipment usually given to the control group at the end of the study. They will then be referred for usual care and will also not be included in the final analysis for the study.
* Unable or unwilling to participate

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Green, MD,MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Group Health Cooperative, Seattle, Washington, United States

REFERENCES:
- [Derived] Green BB, Anderson ML, Cook AJ, Catz S, Fishman PA, McClure JB, Reid RJ. e-Care for heart wellness: a feasibility trial to decrease blood pressure and cardiovascular risk. Am J Prev Med. 2014 Apr;46(4):368-77. doi: 10.1016/j.amepre.2013.11.009. PMID 24650839
- [Derived] Green BB, Anderson ML, Cook AJ, Catz S, Fishman PA, McClure JB, Reid R. Using body mass index data in the electronic health record to calculate cardiovascular risk. Am J Prev Med. 2012 Apr;42(4):342-7. doi: 10.1016/j.amepre.2011.12.009. PMID 22424246